CLINICAL TRIAL: NCT03691779
Title: A Phase 3 Study Evaluating the Pharmacokinetics, Safety, and Tolerability of VX-445/TEZ/IVA Triple Combination Therapy in Cystic Fibrosis Subjects 6 Through 11 Years of Age
Brief Title: Evaluation of VX 445/TEZ/IVA in Cystic Fibrosis Subjects 6 Through 11 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX18-445-106; 2018-001695-38 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: ELX/TEZ/IVA (Experimental): Participants in Part A received ELX 100 milligrams (mg) once daily (qd)/TEZ 50 mg qd/IVA 75 mg every 12 hours (q12h) in the treatment period for 15 days.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA
- Part B: ELX/TEZ/IVA (Experimental): Participants in Part B weighing less than (<) 30 kilograms (kg) at Day 1 received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h and participants weighing greater than equals to (>=) 30 kg at Day 1 received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination tablet orally once daily in the morning.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — IVA tablet orally once daily in the evening.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, tolerability, efficacy, and pharmacodynamic effect of VX-445, tezacaftor (TEZ), and ivacaftor (IVA) when dosed in triple combination (TC) in Cystic Fibrosis (CF) subjects 6 through 11 years of age with F/F and F/MF genotypes.

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous or heterozygous for F508del mutation (F/F or F/MF genotypes)
* Forced expiratory volume in 1 second (FEV1) value ≥40% of predicted mean for age, sex, and height.

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status.
* Solid organ or hematological transplantation.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia's Children's Hospital, Vancouver
- Ireland (2):
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Temple Street, Dublin
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Zemanick ET, Taylor-Cousar JL, Davies J, Gibson RL, Mall MA, McKone EF, McNally P, Ramsey BW, Rayment JH, Rowe SM, Tullis E, Ahluwalia N, Chu C, Ho T, Moskowitz SM, Noel S, Tian S, Waltz D, Weinstock TG, Xuan F, Wainwright CE, McColley SA. A Phase 3 Open-Label Study of Elexacaftor/Tezacaftor/Ivacaftor in Children 6 through 11 Years of Age with Cystic Fibrosis and at Least One F508del Allele. Am J Respir Crit Care Med. 2021 Jun 15;203(12):1522-1532. doi: 10.1164/rccm.202102-0509OC. PMID 33734030
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts, Part A and Part B. All results were planned to be analyzed and reported separately for Part A and Part B of the study.
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants 6 through 11 years of age who were homozygous for F508del (F/F) genotype or heterozygous for F508del and a CF transmembrane conductance regulator gene (CFTR) minimal function mutation (F/MF) genotypes.
Groups:
- Part A: ELX/TEZ/IVA: Participants in Part A received elexacaftor (ELX) 100 milligrams (mg) once daily (qd)/tezacaftor (TEZ) 50 mg qd/ivacaftor (IVA) 75 mg every 12 hours (q12h) in the treatment period for 15 days.
Period: Part A (15 Days)
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
Started | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Part B (24 Weeks)
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
Started | 0 | 66 (Out of the 16 participants from Part A, 11 participants also participated in Part B of the study.)
Completed | 0 | 64
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of consent (not due to AE) | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population included all enrolled participants who carry the intended CFTR allele mutation and received at least 1 dose of study drug in the respective part of the study.
Groups:
- ELX/TEZ/IVA: Part A: Participants in Part A received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h in the treatment period for 15 days.
  Part B: Participants in Part B weighing <30 kg at Day 1 received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h and participants weighing >=30 kg at Day 1 received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants] — Population: Data were planned to be analyzed and reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (15 Days): number analyzed (Participants) | 16
    Part A (15 Days): <=18 years | 16
    Part A (15 Days): Between 18 and 65 years | 0
    Part A (15 Days): >=65 years | 0
    Part B (24 Weeks): number analyzed (Participants) | 66
    Part B (24 Weeks): <=18 years | 66
    Part B (24 Weeks): Between 18 and 65 years | 0
    Part B (24 Weeks): >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were planned to be analyzed and reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (15 Days): number analyzed (Participants) | 16
    Part A (15 Days): Female | 11
    Part A (15 Days): Male | 5
    Part B (24 Weeks): number analyzed (Participants) | 66
    Part B (24 Weeks): Female | 39
    Part B (24 Weeks): Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were planned to be analyzed and reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (15 Days): number analyzed (Participants) | 16
    Part A (15 Days): Hispanic or Latino | 0
    Part A (15 Days): Not Hispanic or Latino | 16
    Part A (15 Days): Unknown or Not Reported | 0
    Part B (24 Weeks): number analyzed (Participants) | 66
    Part B (24 Weeks): Hispanic or Latino | 0
    Part B (24 Weeks): Not Hispanic or Latino | 58
    Part B (24 Weeks): Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were planned to be analyzed and reported separately for Part A and Part B of the study. Here "number analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A (15 Days): number analyzed (Participants) | 16
    Part A (15 Days): American Indian or Alaska Native | 0
    Part A (15 Days): Asian | 0
    Part A (15 Days): Native Hawaiian or Other Pacific Islander | 0
    Part A (15 Days): Black or African American | 0
    Part A (15 Days): White | 16
    Part A (15 Days): More than one race | 0
    Part A (15 Days): Unknown or Not Reported | 0
    Part B (24 Weeks): number analyzed (Participants) | 66
    Part B (24 Weeks): American Indian or Alaska Native | 0
    Part B (24 Weeks): Asian | 0
    Part B (24 Weeks): Native Hawaiian or Other Pacific Islander | 0
    Part B (24 Weeks): Black or African American | 0
    Part B (24 Weeks): White | 57
    Part B (24 Weeks): More than one race | 1
    Part B (24 Weeks): Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of ELX, TEZ, and IVA
Time Frame: Part A: Day 15
Population: Pharmacokinetic (PK) set for Part A included all participants who have received at least 1 dose of study drug in Part A. Here, the "number analyzed" signifies participants who were evaluable at the specified time point. This outcome measure was planned only for Part A arm.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Groups:
- Part A: ELX/TEZ/IVA: Participants in Part A received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h in the treatment period for 15 days.
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
microgram per milliliter (mcg/mL)
  ELX: number analyzed (Participants) | 15
  ELX | 6.13 (1.52)
  TEZ: number analyzed (Participants) | 15
  TEZ | 6.93 (1.96)
  IVA: number analyzed (Participants) | 15
  IVA | 1.01 (0.281)

2. Primary Outcome: Part A: Observed Pre-dose Plasma Concentration (Ctrough) of ELX, TEZ, and IVA
Time Frame: Part A: Day 15
Population: PK set (Part A). Here, the "number analyzed" signifies participants who were evaluable at the specified time point. This outcome measure was planned only for Part A arm.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  ELX: number analyzed (Participants) | 15
  ELX | 2.86 (1.37)
  TEZ: number analyzed (Participants) | 15
  TEZ | 1.06 (0.366)
  IVA: number analyzed (Participants) | 15
  IVA | 0.297 (0.173)

3. Primary Outcome: Part A: Area Under the Concentration Versus Time Curve From 0 to 24 Hours (AUC0-24h) of ELX, TEZ, and IVA
Time Frame: Part A: Day 15
Population: PK set (Part A). This outcome measure was planned only for Part A arm.
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
hour*microgram per milliliter (h*mcg/mL)
  ELX | 107 (28.7)
  TEZ | 58.4 (13.5)
  IVA | 8.12 (2.93)

4. Primary Outcome: Part B: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Part B: Day 1 Through Safety Follow-up Visit (up to Week 28)
Population: Safety set for Part B included all participants who received at least 1 dose of study drug in Part B. The safety and tolerability analysis for Part B was assessed for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Number; unit: participants
Groups:
- Part B: ELX/TEZ/IVA: Participants in Part B weighing <30 kg at Day 1 received ELX 100 mg qd/TEZ 50 mg qd/IVA 75 mg q12h and participants weighing >=30 kg at Day 1 received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
participants
  Participants With TEAEs | 65
  Participants With SAEs | 1

5. Secondary Outcome: Part A: Cmax of ELX Metabolite (M23-ELX), TEZ Metabolite (M1-TEZ), and IVA Metabolite (M1-IVA)
Time Frame: Part A: Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  M23-ELX: number analyzed (Participants) | 15
  M23-ELX | 1.60 (0.657)
  M1-TEZ: number analyzed (Participants) | 15
  M1-TEZ | 6.26 (1.54)
  M1-IVA: number analyzed (Participants) | 15
  M1-IVA | 2.36 (0.694)

6. Secondary Outcome: Part A: Ctrough of ELX Metabolite (M23-ELX), TEZ Metabolite (M1-TEZ), and IVA Metabolite (M1-IVA)
Time Frame: Part A: Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
mcg/mL
  M23-ELX: number analyzed (Participants) | 15
  M23-ELX | 1.30 (0.585)
  M1-TEZ: number analyzed (Participants) | 15
  M1-TEZ | 4.64 (1.36)
  M1-IVA: number analyzed (Participants) | 15
  M1-IVA | 0.890 (0.460)

7. Secondary Outcome: Part A: AUC0-24h of ELX Metabolite (M23-ELX) and TEZ Metabolite (M1-TEZ)
Time Frame: Part A: Day 15
Population: PK set (Part A). This outcome measure was planned only for Part A arm.
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
h*mcg/mL
  M23-ELX | 35.6 (13.2)
  M1-TEZ | 133 (30.4)

8. Secondary Outcome: Part A: Area Under the Concentration Versus Time Curve From 0 to 6 Hours (AUC0-6h) of IVA Metabolite (M1-IVA)
Description: The AUC data was analyzed for up to 6 hours for IVA metabolite (M1-IVA). Therefore, AUC0-6h is reported for M1-IVA metabolite.
Time Frame: Part A: Day 15
Population: PK set (Part A). Here "overall number of participants analyzed" signifies participants who were evaluable at the specified time points. This outcome measure was planned only for Part A arm.
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 15
h*mcg/mL | 9.41 (3.06)

9. Secondary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With TEAEs and SAEs
Time Frame: Part A: Day 1 Through Safety Follow-up Visit (up to Day 43)
Population: Safety set for Part A included all participants who received at least 1 dose of study drug in Part A. This outcome measure was planned only for Part A arm.
Measure: Number; unit: participants
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 16
participants
  Participants With TEAEs | 12
  Participants With SAEs | 0

10. Secondary Outcome: Part B: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Part B: From Baseline Through Week 24
Population: Full analysis set (FAS) for Part B included all enrolled participants who carry the intended CFTR allele mutation and received at least 1 dose of study drug in Part B. The efficacy analysis for Part B was assessed for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
percentage points | 10.2 [7.9 to 12.6]

11. Secondary Outcome: Part B: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: Part B: From Baseline Through Week 24
Population: FAS (Part B). The efficacy analysis for Part B was assessed for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
millimole per liter (mmol/L) | -60.9 [-63.7 to -58.2]

12. Secondary Outcome: Part B: Absolute Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Part B: From Baseline Through Week 24
Population: FAS (Part B). The efficacy analysis for Part B was planned for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
units on a scale | 7.0 [4.7 to 9.2]

13. Secondary Outcome: Part B: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kg divided by squared height in meters (m^2).
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
kg/m^2 | 1.02 [0.76 to 1.28]

14. Secondary Outcome: Part B: Absolute Change in BMI For-Age Z-Score
Description: BMI was defined as weight in kg divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
z-score | 0.37 [0.26 to 0.48]

15. Secondary Outcome: Part B: Absolute Change in Weight
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
kg | 3.0 [2.5 to 3.5]

16. Secondary Outcome: Part B: Absolute Change in Weight-for-age Z-Score
Description: The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
z-score | 0.25 [0.16 to 0.33]

17. Secondary Outcome: Part B: Absolute Change in Height
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters (cm)
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
centimeters (cm) | 2.3 [1.9 to 2.7]

18. Secondary Outcome: Part B: Absolute Change in Height-for-Age Z-Score
Description: as for outcome 16
Time Frame: Part B: From Baseline at Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
z-score | -0.05 [-0.12 to 0.01]

19. Secondary Outcome: Part B: Drug Acceptability Assessment Using Modified Facial Hedonic Scale
Description: The study drug acceptability (participant reaction) was assessed by a visual analog scale that incorporates a 5 point facial hedonic scale (Liked it Very Much, Liked it a Little, Not sure, Disliked it a Little, Disliked it Very Much). Number of participants with the indicated categorical response in the drug acceptability assessment were reported.
Time Frame: Part B: At Week 24
Population: FAS (Part B). The efficacy analysis for Part B was assessed for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 33
participants
  Liked it Very Much | 16
  Liked it a Little | 6
  Not sure | 10
  Disliked it a Little | 1
  Disliked it Very Much | 0

20. Secondary Outcome: Part B: Number of Pulmonary Exacerbations Events
Description: Pulmonary exacerbation was defined as new or changed treatment with oral, inhaled, or intravenous antibiotics and fulfillment of pre-specified protocol defined criteria. The total number of pulmonary exacerbations events across all participants were reported.
Time Frame: Part B: From Baseline Through Week 24
Population: as for outcome 11
Measure: Number; unit: pulmonary exacerbations events
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
pulmonary exacerbations events | 4

21. Secondary Outcome: Part B: Number of CF Related Hospitalizations
Description: The total number of CF related hospitalization events across all participants were reported.
Time Frame: Part B: From Baseline Through Week 24
Population: as for outcome 11
Measure: Number; unit: hospitalizations
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
hospitalizations | 0

22. Secondary Outcome: Part B: Ctrough of ELX, ELX Metabolite (M23-ELX), TEZ, TEZ Metabolite (M1-TEZ), IVA and IVA Metabolite (M1-IVA)
Time Frame: Part B: At Week 4
Population: The PK set for Part B included all participants who have received at least 1 dose of study drug in Part B. Here "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 65
mcg/mL
  ELX: Week 4 (<30 kg): number analyzed (Participants) | 33
  ELX: Week 4 (<30 kg) | 2.71 (1.77)
  ELX: Week 4 (>=30 kg): number analyzed (Participants) | 30
  ELX: Week 4 (>=30 kg) | 5.69 (3.00)
  M23-ELX: Week 4 (<30 kg): number analyzed (Participants) | 33
  M23-ELX: Week 4 (<30 kg) | 1.59 (1.24)
  M23-ELX: Week 4 (>=30 kg): number analyzed (Participants) | 30
  M23-ELX: Week 4 (>=30 kg) | 4.41 (2.97)
  TEZ: Week 4 (<30 kg): number analyzed (Participants) | 33
  TEZ: Week 4 (<30 kg) | 1.43 (1.19)
  TEZ: Week 4 (>=30 kg): number analyzed (Participants) | 30
  TEZ: Week 4 (>=30 kg) | 2.37 (1.07)
  M1-TEZ: Week 4 (<30 kg): number analyzed (Participants) | 33
  M1-TEZ: Week 4 (<30 kg) | 5.57 (1.78)
  M1-TEZ: Week 4 (>=30 kg): number analyzed (Participants) | 30
  M1-TEZ: Week 4 (>=30 kg) | 8.12 (1.88)
  IVA: Week 4 (<30 kg): number analyzed (Participants) | 33
  IVA: Week 4 (<30 kg) | 0.455 (0.681)
  IVA: Week 4 (>=30 kg): number analyzed (Participants) | 30
  IVA: Week 4 (>=30 kg) | 0.851 (0.489)
  M1-IVA: Week 4 (<30 kg): number analyzed (Participants) | 33
  M1-IVA: Week 4 (<30 kg) | 1.00 (0.630)
  M1-IVA: Week 4 (>=30 kg): number analyzed (Participants) | 30
  M1-IVA: Week 4 (>=30 kg) | 2.18 (1.04)

23. Secondary Outcome: Part B: Absolute Change in Lung Clearance Index 2.5 (LCI2.5)
Description: LCI 2.5 represents the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting value.
Time Frame: Part B: From Baseline Through Week 24
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: lung clearance index
Arm/Group | Part B: ELX/TEZ/IVA
Number analyzed (Participants) | 66
lung clearance index | -1.71 [-2.11 to -1.30]

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (up to Day 43 for Part A, up to Week 28 for Part B)
Description: The safety analysis for Part B was assessed for the overall treatment arm, irrespective of weight based dose regimen. Therefore, the analysis is reported for the single triple combination (Part B: ELX/TEZ/IVA) arm. MedDRA version 21.1 applied for Part A, MedDRA version 23.0 applied for Part B.
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/66
Other Adverse Events (participants affected / at risk) | 12/16 | 62/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=16) | Part B: ELX/TEZ/IVA (N=66)
Metapneumovirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=16) | Part B: ELX/TEZ/IVA (N=66)
Abdominal pain (Gastrointestinal disorders) | 1 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 7
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 7
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 5
Pyrexia (General disorders) | 1 | 14
Vessel puncture site pain (General disorders) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 0 | 7
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 11
Viral upper respiratory tract infection (Infections and infestations) | 0 | 8
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Human rhinovirus test positive (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 16
Lethargy (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 28
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT03691779/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03691779/SAP_001.pdf